CLINICAL TRIAL: NCT00713999
Title: Study of Reproductive Health in Rural Madagascar With Emphasis on Urogenital Schistosomiasis and Sexually Transmitted Infections
Brief Title: Urogenital Schistosomiasis and Sexually Transmitted Infections in Madagascar
Acronym: FGS/MGS/STI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Peter Derek Christian Leutscher, MD,PhD, Danish Bilharziasis Laboratory
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IPM/DBL 01; RFU 1008600437
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2008-07-14 (Estimated); Status verified 2008-07

CONDITIONS: Sexually Transmitted Infections; Schistosoma Haematobium
Keywords: Sexually transmitted infections; Urogenital schistosomiasis; Schistosoma haematobium; Reproductive health; Pelvic examination; Ultrasonography; Questionnaire; Madagascar
MeSH Terms: conditions — Sexually Transmitted Diseases; Schistosomiasis haematobia | interventions — Therapeutics; Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- STI/PZQ 1 (Experimental): Baseline and post-treatment follow-up (anti-STI and praziquantel Rx)
  Interventions: Drug: Treatment with anti-STI and anti-schistosoma regimens

INTERVENTIONS:
Drug: Treatment with anti-STI and anti-schistosoma regimens — Anti-STI regimen: ciprofloxacin 500mg orally, doxycycline 100mg BID orally 7 days and metronidazole 2g orally (cefuroxime im and/or azithromycin alternatively for pregnant and breastfeeding women) Anti-schistosoma regimen: Praziquantel 40mg/kg
  Other Names: Biltricide

SUMMARY:
A cross-sectional study of urogenital schistosomiasis and sexually transmitted infections (STI) prevalence and associated morbidity in a rural community in Madagascar. Clearance of infections and resolution of morbidity were subsequently studied in two phases following systematic anti-STI and anti-schistosoma treatment, respectively.

DETAILED DESCRIPTION:
The study was conducted in the Schistosoma haematobium high-endemic SIRAMA sugarcane plantation near the Ambilobe town in the northern province of Diego Suarez in Madagascar. A neighboring low-endemic village, Mataipako, was selected a control village. Participants aged 15 to 49 years old from SIRAMA were included in the study if positive for S.haematobium egg in urine.

A questionnaire addressing previous medical history and current urogenital symptoms was applied. A physical examination, including ultrasonophical (US) examination of urinary tract by transabdominal route, was undertaken. A pelvic examination, including transvaginal US was performed in women. In men, the prostate and the seminal vesicles were examined by transrectal US.

The following sexually transmitted infections (STI) were systematically assessed:

* Neisseria gonorrheae
* Chlamydia trachomatis
* Mycoplasma genitalium
* Trichomonas
* Treponema pallidum
* Herpes simplex 1 and 2

After baseline assessment, all participants (and partners) were systematically treated with an anti-STI regimen according to the existing guidelines by the Ministry of Health in Madagascar.

Re-assessment by questionnaire, physical examination and sampling for STIs was undertaken 4 weeks later followed by systematic praziquantel treatment to general community, including study participants.

A final follow-up study following the baseline protocol was conducted 5 months later.

ELIGIBILITY:
Inclusion Criteria:

* adults
* positive Schistosoma haematobium egg excretion in urine
* signed written consensus

Exclusion Criteria:

* children
* negative Schistosoma haematobium egg excretion in urine

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 680 (Actual)
Dates: Start 2001-08; Primary Completion 2002-04 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Measurement of urogenital schistosomiasis and STI prevalence | 2 months

SECONDARY OUTCOMES:
Urogenital and STI associated morbidity | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter DC Leutscher, MD, PhD, Principal Investigator — Danish Bilharziasis Laboratory
Locations (1):
- Institut Pasteur, Antananarivo, Madagascar